CLINICAL TRIAL: NCT00768079
Title: A Phase 2, Multicenter, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of Intravenously Administered MEDI-563, A Humanized Anti-interleukin-5 Receptor Alpha Monoclonal Antibody, on Asthma Control Following Acute Exacerbations in Adults
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of Intravenously Administered Benralizumab (MEDI-563).
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MI-CP186
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2020-10-12 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-10

CONDITIONS: Asthma
Keywords: Benralizumab; MEDI-563; Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): A single dose of placebo matched to benralizumab (MEDI-563) intravenous infusion over at least 30 minutes on Day 0.
  Interventions: Other: Placebo
- Benralizumab 0.3 mg/kg (Experimental): A single dose of benralizumab (MEDI-563) 0.3 milligram per kilogram (mg/kg) of body weight intravenous infusion over at least 30 minutes on Day 0.
  Interventions: Biological: Benralizumab
- Benralizumab 1.0 mg/kg (Experimental): A single dose of benralizumab (MEDI-563) 1.0 mg/kg of body weight intravenous infusion over at least 30 minutes on Day 0.
  Interventions: Biological: Benralizumab

INTERVENTIONS:
Other: Placebo — A single dose of placebo matched to benralizumab (MEDI-563) intravenous infusion over at least 30 minutes on Day 0.
  Arms: Placebo
Biological: Benralizumab — A single dose of benralizumab (MEDI-563) 0.3 or 1 mg/kg of body weight intravenous infusion over at least 30 minutes on Day 0.
  Other Names: MEDI-563
  Arms: Benralizumab 0.3 mg/kg; Benralizumab 1.0 mg/kg

SUMMARY:
The study will evaluate the effect of two intravenous dose regimens of benralizumab (MEDI-563) on the proportion of adult subjects with asthma exacerbations who required an urgent healthcare visit for treatment of an acute asthma exacerbation.

DETAILED DESCRIPTION:
The study will evaluate the effect of two intravenous dose regimens of benralizumab (MEDI-563) (0.3 milligram per kilogram [mg/kg] of body weight and 1.0 mg/kg of body weight) on the proportion of adult subjects with asthma exacerbations (relapse and de novo) who required an urgent healthcare visit for treatment of an acute asthma exacerbation.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged 18 to 60 years at the time of the administration of investigational product
* Written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization (applies to covered entities in the US only) obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations
* Physician-diagnosed asthma with a duration of greater than or equal to (>=) 2 years by medical chart or subject report
* Had an asthma exacerbation requiring urgent care in the year prior to screening
* Meets National Heart, Lung, and Blood Institute (NHLBI) for persistent asthma in the 3 months prior to the current urgent healthcare visit
* Current asthma exacerbation that must have lasted >= 2 hours prior to arrival to the urgent healthcare setting
* Requires at least 2 treatments of inhaled bronchodilators for the current asthma exacerbation in the urgent healthcare setting or within the emergency medical system (EMS) for >= 1 hour
* Shows an FEV1 or PEF of not more than 70 percent (%) predicted after 1 hour of treatment of the current asthma exacerbation
* Women of child-bearing potential, unless surgically sterile (including tubal ligation) and/or at least 2 years post-menopausal, must have used 2 effective methods of avoiding pregnancy (including oral, transdermal, or implanted contraceptives, intrauterine device, female condom with spermicide, diaphragm with spermicide, cervical cap, abstinence, use of a condom with spermicide by the sexual partner, or sterile sexual partner) from screening through the end of the study (Day 84; Cessation of birth control after this point should be discussed with a responsible physician)
* Men, unless surgically sterile, must likewise practice 2 effective methods of birth control (condom with spermicide or abstinence) and must use such precautions from Day 0 through Day 84
* Otherwise healthy by medical history and physical examination
* A chest x-ray that is normal for an asthmatic population and excludes alternative diagnosis per the investigation
* Ability to complete the follow-up period until Day 168 as required by protocol
* The investigator has determined that the subject is clinically stable and the FEV1, is >= 30% predicted prior to receiving investigational product on Day 0.

Exclusion Criteria:

* Known history of allergy or reaction to any component of the investigational product formulation
* Acute illness other than asthma at the start of the study
* Fever more than (>) 38.6 degrees Celsius (C) (>101.5 degrees Fahrenheit [F])
* Current acute asthma attack is due to aspirin-induced asthma
* Current asthma episode is an anaphylactoid/anaphylactic reaction presenting with acute bronchospasm
* Evidence of clinically significant non-respiratory active infection, including ongoing chronic infection
* History or current prolonged diarrhea, abdominal pain, and/or blood and mucus in stools or have minor symptoms and have exposure to stream or lake water, been exposed to someone who has a parasitic infection (like a family member), or study subject has traveled outside the United States of America (USA) and/or Canada within the last year
* Use of immunosuppressive medication (except oral prednisone and inhaled and topical corticosteroids) within 30 days before randomization into the study
* Have received Xolair within 6 months before randomization into the study
* Receipt of immunoglobulin or blood products within 30 days before randomization into the study
* Receipt of any investigational drug therapy within 6 months before the first dose of investigational product in this study through Day 168
* History of primary immunodeficiency
* Previous medical history, or evidence, of an intercurrent illness that may compromise the safety of the subject in the study
* History of clinically significant abnormality on ECG in the opinion of the investigator
* Pregnancy (must have a negative serum pregnancy test prior to the first dose of investigational product)
* Breastfeeding or lactating woman
* History of treatment for alcohol or drug abuse within the past year
* Diagnosis of chronic obstructive pulmonary disease (COPD) by a healthcare professional
* Evidence of any clinically significant systemic disease on physical examination
* History of cancer except basal cell carcinoma or in situ carcinoma of the cervix treated with apparent success with curative therapy >1 year prior to entry or other malignancies treated with apparent success with curative therapy >5 years prior to entry
* Known exposure to inhaled occupational agents or fumes with an established diagnosis of occupational asthma
* Any condition (that is, impending ventilatory failure or hemodynamic compromise) that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of study results
* Any employee of the clinical study site who is involved with the conduct of the study
* History of cigarette smoking >20 pack years
* Previously received benralizumab (MEDI-563)
* Asthma exacerbation due to acute inhalational exposure.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2009-02-02 (Actual); Primary Completion 2010-12-17 (Actual); Study Completion 2011-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph M. Parker, M.D., Study Director — MedImmune LLC
Locations (11):
- United States (9):
  - Research Site, Tampa, Florida
  - Research Site, Springfield, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, East Meadow, New York
  - Research Site, New Hyde Park, New York
  - Research Site, Stony Brook, New York
  - Research Site, Greenville, North Carolina
  - Research Site, Cleveland, Ohio
  - Research Site, Providence, Rhode Island
- Canada (2):
  - Research Site, Edmonton, Alberta
  - Research Site, Halifax, Nova Scotia

REFERENCES:
- [Derived] Nowak RM, Parker JM, Silverman RA, Rowe BH, Smithline H, Khan F, Fiening JP, Kim K, Molfino NA. A randomized trial of benralizumab, an antiinterleukin 5 receptor alpha monoclonal antibody, after acute asthma. Am J Emerg Med. 2015 Jan;33(1):14-20. doi: 10.1016/j.ajem.2014.09.036. Epub 2014 Oct 5. PMID 25445859
- See also: MEDI-563_CP-186_Protocol_Redacted_16Dec2014 — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=18&filename=MEDI-563_CP-186_Protocol_Redacted_16Dec2014.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 110 participants were randomized in the study.
Period: Overall Study
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Started | 38 | 36 | 36
Completed | 36 | 35 | 32
Not Completed | 2 | 1 | 4
Not completed — Lost to Follow-up | 2 | 0 | 4
Not completed — Participant incarcerated | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population included all participants who were randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg | Total
Number analyzed (Participants) | 38 | 36 | 36 | 110
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.9 (10.5) | 37.9 (11.4) | 34.8 (10.0) | 36.2 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 24 | 23 | 77
  Male | 8 | 12 | 13 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 2 | 7 | 15
  Not Hispanic or Latino | 32 | 34 | 29 | 95
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 26 | 19 | 19 | 64
  White | 11 | 14 | 16 | 41
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Asthma Exacerbations at Week 12
Description: Percentage of participants who required urgent healthcare visit for treatment of acute asthma exacerbation were reported. As per protocol, asthma exacerbation (relapse/de novo) was defined as either 1) increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) that did not resolve within 2 hours after use of rescue albuterol or corticosteroids and required an unscheduled medical visit or 2) during scheduled study visit, participant had acute worsening of asthma symptoms and a reduction of greater than or equal to (>=) 20 percent (%) in Peak Expiratory Flow (PEF) or Forced Expiratory Volume in 1 Second (FEV1), which in the opinion of the investigator required treatment with systemic corticosteroids. Asthma exacerbations were analyzed in a non-adjudicated manner (by investigator), which were then adjudicated in a blinded fashion by the sponsor medical monitor prior to database lock to determine whether the reported exacerbation met the protocol definition.
Time Frame: Week 12
Population: Evaluable population included all participants who received any study drug and were followed according to the protocol through Day 42.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
percentage of participants
  Non-adjudicated Exacerbations | 38.9 | 25.0 | 41.7
  Adjudicated Exacerbations | 38.9 | 25.0 | 41.7
Statistical Analysis 1: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.312, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.312, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An adverse event (AE) was any untoward medical occurrence attributed to study drug in a participant who received study drug. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between administration of study drug and Day 84 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 0 to Day 84
Population: Safety population included all participants who received any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 38 | 36 | 36
Participants
  TEAEs | 30 | 32 | 30
  TESAEs | 9 | 8 | 11

3. Secondary Outcome: Percentage of Participants With Asthma Exacerbations at Week 4 and Week 24
Description: Percentage of participants who required an urgent healthcare visit for treatment of an acute asthma exacerbation were reported. As per protocol, asthma exacerbation (relapse or de novo) was defined as either 1) an increase of asthma symptoms (cough, wheeze, chest tightness, and/or shortness of breath) that did not resolve within 2 hours after the use of rescue albuterol or corticosteroids and required an unscheduled medical visit or 2) during a scheduled study visit, the participant had acute worsening of asthma symptoms and a reduction of >=20% in PEF or FEV1, which in the opinion of the investigator required treatment with systemic corticosteroids. Asthma exacerbations were analyzed in a non-adjudicated manner (by investigator), which were then adjudicated in a blinded fashion by the sponsor medical monitor prior to database lock to determine whether the reported exacerbation met the protocol definition.
Time Frame: Weeks 4 and 24
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
percentage of participants
  Week 4: Non-adjudicated Exacerbations | 22.2 | 11.1 | 22.2
  Week 4: Adjudicated Exacerbations | 22.2 | 11.1 | 22.2
  Week 24: Non-adjudicated Exacerbations | 47.2 | 36.1 | 50.0
  Week 24: Adjudicated Exacerbations | 47.2 | 36.1 | 50.0
Statistical Analysis 1: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Week 4, non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.343, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Week 4, non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Week 4, adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.343, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Week 4, adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 5: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Week 24, non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.474, Fisher Exact
Statistical Analysis 6: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Week 24, non-adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact
Statistical Analysis 7: Comparison: Placebo vs Benralizumab 0.3 mg/kg; Week 24, adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 0.474, Fisher Exact
Statistical Analysis 8: Comparison: Placebo vs Benralizumab 1.0 mg/kg; Week 24, adjudicated exacerbations: Fisher's exact test was used for statistical analysis; Test type: Superiority or Other; p = 1.000, Fisher Exact

4. Secondary Outcome: Asthma Control Questionnaire (ACQ) Scores
Description: Asthma Control Questionnaire (ACQ) is a participant-reported questionnaire to assess the asthma control with 6 items assessing night-time waking, symptoms on waking, activity limitation, shortness of breath, wheeze, and rescue short-acting beta agonist use. Each item was rated on a 7-point Likert scale ranging from 0 (no impairment) to 6 (maximum impairment). Overall ACQ score is the mean of the 6 item scores with a score range of 0 (well controlled) to 6 (extremely poor controlled). Results were reported for overall ACQ score and 6 item scores.
Time Frame: Days 0, 7, 42, and 84
Population: Evaluable population included all participants who received any study drug and were followed according to the protocol through Day 42. Here, "Number Analyzed" signified those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Overall ACQ: Day 0 | 3.69 (0.82) | 3.72 (1.18) | 3.26 (1.27)
  Overall ACQ: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Overall ACQ: Day 7 | 1.89 (1.16) | 1.89 (1.36) | 1.52 (0.96)
  Overall ACQ: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Overall ACQ: Day 42 | 1.70 (1.23) | 1.76 (1.25) | 1.50 (1.13)
  Overall ACQ: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Overall ACQ: Day 84 | 1.59 (1.23) | 1.75 (1.33) | 1.70 (1.12)
  Night-time waking: Day 0 | 3.1 (1.4) | 3.5 (1.8) | 2.9 (1.7)
  Night-time waking: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Night-time waking: Day 7 | 1.7 (1.6) | 1.7 (1.7) | 1.0 (1.0)
  Night-time waking: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Night-time waking: Day 42 | 1.4 (1.6) | 1.6 (1.5) | 1.2 (1.4)
  Night-time waking: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Night-time waking: Day 84 | 1.3 (1.4) | 1.4 (1.6) | 1.2 (1.2)
  Symptoms on waking: Day 0 | 3.4 (1.4) | 3.5 (1.5) | 2.8 (1.5)
  Symptoms on waking: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Symptoms on waking: Day 7 | 1.8 (1.3) | 2.0 (1.4) | 1.4 (1.2)
  Symptoms on waking: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Symptoms on waking: Day 42 | 1.6 (1.3) | 1.6 (1.3) | 1.2 (1.0)
  Symptoms on waking: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Symptoms on waking: Day 84 | 1.5 (1.6) | 1.7 (1.4) | 1.6 (1.2)
  Activity limitation: Day 0 | 3.6 (1.3) | 3.5 (1.4) | 3.2 (1.8)
  Activity limitation: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Activity limitation: Day 7 | 1.7 (1.3) | 1.8 (1.5) | 1.5 (1.5)
  Activity limitation: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Activity limitation: Day 42 | 1.6 (1.5) | 1.6 (1.5) | 1.4 (1.3)
  Activity limitation: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Activity limitation: Day 84 | 1.3 (1.3) | 1.5 (1.3) | 2.0 (1.9)
  Shortness of breath: Day 0 | 4.4 (1.0) | 4.2 (1.3) | 3.7 (1.5)
  Shortness of breath: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Shortness of breath: Day 7 | 1.9 (1.4) | 2.1 (1.5) | 1.8 (1.4)
  Shortness of breath: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Shortness of breath: Day 42 | 2.0 (1.3) | 2.1 (1.5) | 1.9 (1.5)
  Shortness of breath: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Shortness of breath: Day 84 | 1.8 (1.3) | 2.0 (1.4) | 1.9 (1.4)
  Wheeze: Day 0 | 4.5 (1.1) | 4.2 (1.5) | 4.0 (1.6)
  Wheeze: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Wheeze: Day 7 | 2.6 (1.9) | 2.2 (1.6) | 2.0 (1.8)
  Wheeze: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Wheeze: Day 42 | 2.1 (1.5) | 2.0 (1.5) | 1.8 (1.5)
  Wheeze: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Wheeze: Day 84 | 2.1 (1.7) | 2.2 (1.7) | 1.8 (1.6)
  Rescue beta-2 agonist use: Day 0 | 3.0 (1.3) | 3.3 (1.6) | 3.2 (1.5)
  Rescue beta-2 agonist use: Day 7: number analyzed (Participants) | 36 | 36 | 35
  Rescue beta-2 agonist use: Day 7 | 1.7 (1.1) | 1.6 (1.5) | 1.3 (0.9)
  Rescue beta-2 agonist use: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Rescue beta-2 agonist use: Day 42 | 1.5 (1.3) | 1.6 (1.3) | 1.6 (1.6)
  Rescue beta-2 agonist use: Day 84: number analyzed (Participants) | 36 | 35 | 32
  Rescue beta-2 agonist use: Day 84 | 1.5 (1.2) | 1.7 (1.4) | 1.8 (1.3)

5. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Recorded at Study Sites
Description: The FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Spirometry was performed with the participant in the sitting position at study sites by the investigator or qualified designee according to American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines. Multiple forced expiratory efforts (at least 2 but no more than 5) were performed for each office spirometry session and the 2 best efforts that met ATS/ERS acceptability and reproducibility criteria were recorded. The best efforts were based on the highest FEV1. The maximum FEV1 of the 2 best efforts was used for the analysis.
Time Frame: Days 0, 7, 42, and 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
liters
  Day 0: number analyzed (Participants) | 36 | 35 | 34
  Day 0 | 1.696 (0.523) | 1.689 (0.698) | 2.067 (0.746)
  Day 7: number analyzed (Participants) | 36 | 35 | 35
  Day 7 | 2.008 (0.632) | 2.003 (0.655) | 2.254 (0.723)
  Day 42: number analyzed (Participants) | 33 | 35 | 34
  Day 42 | 1.962 (0.714) | 2.130 (0.713) | 2.150 (0.723)
  Day 84: number analyzed (Participants) | 36 | 35 | 32
  Day 84 | 2.048 (0.761) | 2.043 (0.710) | 2.209 (0.791)

6. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) Recorded at Home
Description: The FEV1 is the maximal volume of air exhaled in the first second of a forced expiration from a position of full inspiration. Home peak flow testing for FEV1 was performed every morning while sitting or standing prior to using any medication (if needed) for asthma. Mean FEV1 values for each week were reported starting from Day 1 to Day 84.
Time Frame: Day 1 to Day 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
liters
  Day 1 to 7: number analyzed (Participants) | 34 | 32 | 33
  Day 1 to 7 | 1.6346 (0.4868) | 1.7119 (0.6309) | 1.8404 (0.7222)
  Day 8 to 14: number analyzed (Participants) | 31 | 29 | 33
  Day 8 to 14 | 1.7800 (0.5608) | 1.8562 (0.6467) | 1.7674 (0.7305)
  Day 15 to 21: number analyzed (Participants) | 31 | 31 | 30
  Day 15 to 21 | 1.7024 (0.5200) | 1.7874 (0.6529) | 1.8219 (0.7241)
  Day 22 to 28: number analyzed (Participants) | 30 | 31 | 30
  Day 22 to 28 | 1.6751 (0.5814) | 1.8188 (0.6461) | 1.8351 (0.7107)
  Day 29 to 35: number analyzed (Participants) | 31 | 32 | 31
  Day 29 to 35 | 1.6446 (0.4962) | 1.7937 (0.6229) | 1.7486 (0.7093)
  Day 36 to 42: number analyzed (Participants) | 32 | 30 | 31
  Day 36 to 42 | 1.7230 (0.5844) | 1.7935 (0.6341) | 1.7298 (0.6923)
  Day 43 to 49: number analyzed (Participants) | 33 | 31 | 28
  Day 43 to 49 | 1.7326 (0.5426) | 1.7999 (0.6735) | 1.7803 (0.6655)
  Day 50 to 56: number analyzed (Participants) | 33 | 30 | 28
  Day 50 to 56 | 1.6965 (0.5756) | 1.7532 (0.6530) | 1.7806 (0.6558)
  Day 57 to 63: number analyzed (Participants) | 32 | 29 | 30
  Day 57 to 63 | 1.6600 (0.6013) | 1.7682 (0.6619) | 1.8504 (0.7636)
  Day 64 to 70: number analyzed (Participants) | 30 | 30 | 30
  Day 64 to 70 | 1.7218 (0.6308) | 1.8735 (0.7701) | 1.7904 (0.7959)
  Day 71 to 77: number analyzed (Participants) | 28 | 27 | 30
  Day 71 to 77 | 1.7180 (0.5969) | 1.7811 (0.6721) | 1.7401 (0.6891)
  Day 78 to 84: number analyzed (Participants) | 29 | 30 | 31
  Day 78 to 84 | 1.7591 (0.6944) | 1.6655 (0.6032) | 1.7818 (0.7009)

7. Secondary Outcome: Peak Expiratory Flow (PEF) Recorded at Home
Description: The PEF is a participant's maximum speed of expiration, as measured with a peak flow meter. Home peak flow testing for PEF was performed every morning while sitting or standing prior to using any medication (if needed) for asthma. Mean PEF values for each week were reported starting from Day 1 to Day 84.
Time Frame: Day 1 to Day 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: liters per minute (L/min)
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
liters per minute (L/min)
  Day 1 to 7: number analyzed (Participants) | 34 | 32 | 33
  Day 1 to 7 | 161.845 (45.186) | 179.000 (61.653) | 177.929 (58.791)
  Day 8 to 14: number analyzed (Participants) | 31 | 29 | 33
  Day 8 to 14 | 175.093 (50.914) | 186.538 (52.945) | 172.811 (59.941)
  Day 15 to 21: number analyzed (Participants) | 31 | 31 | 30
  Day 15 to 21 | 169.489 (51.560) | 180.627 (55.853) | 180.362 (60.894)
  Day 22 to 28: number analyzed (Participants) | 30 | 31 | 30
  Day 22 to 28 | 163.844 (57.753) | 183.066 (54.902) | 181.199 (62.497)
  Day 29 to 35: number analyzed (Participants) | 31 | 32 | 31
  Day 29 to 35 | 163.999 (53.078) | 179.064 (55.297) | 171.458 (65.889)
  Day 36 to 42: number analyzed (Participants) | 32 | 30 | 31
  Day 36 to 42 | 169.510 (57.745) | 178.373 (51.881) | 168.228 (64.673)
  Day 43 to 49: number analyzed (Participants) | 33 | 31 | 28
  Day 43 to 49 | 171.373 (56.824) | 185.847 (57.767) | 169.727 (65.110)
  Day 50 to 56: number analyzed (Participants) | 33 | 30 | 28
  Day 50 to 56 | 169.487 (58.325) | 178.070 (57.414) | 169.230 (62.696)
  Day 57 to 63: number analyzed (Participants) | 32 | 29 | 30
  Day 57 to 63 | 169.723 (61.318) | 176.761 (56.410) | 169.374 (70.249)
  Day 64 to 70: number analyzed (Participants) | 30 | 30 | 30
  Day 64 to 70 | 166.968 (57.401) | 188.805 (59.186) | 164.368 (66.619)
  Day 71 to 77: number analyzed (Participants) | 28 | 27 | 30
  Day 71 to 77 | 160.717 (61.017) | 175.379 (59.158) | 160.167 (59.618)
  Day 78 to 84: number analyzed (Participants) | 29 | 30 | 31
  Day 78 to 84 | 167.197 (58.690) | 172.788 (56.722) | 164.982 (60.271)

8. Secondary Outcome: Number of Puffs of Rescue Beta-2 Agonist Per Week
Description: Rescue beta-2 agonist use (total number of puffs for the prior day) was collected daily in the morning by the participants in the electronic daily diary provided to them. Participants were instructed not to collect rescue beta-2 agonist used prior to exercise. Average values for each week were reported starting from Day 1 to Day 84.
Time Frame: Day 1 to Day 84
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: puffs per week
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
puffs per week
  Day 1 to 7: number analyzed (Participants) | 34 | 32 | 33
  Day 1 to 7 | 1.95 (1.75) | 1.74 (2.05) | 1.47 (1.76)
  Day 8 to 14: number analyzed (Participants) | 31 | 29 | 33
  Day 8 to 14 | 1.80 (2.01) | 1.63 (1.90) | 1.38 (2.07)
  Day 15 to 21: number analyzed (Participants) | 31 | 31 | 30
  Day 15 to 21 | 1.57 (2.00) | 2.01 (3.34) | 1.42 (1.70)
  Day 22 to 28: number analyzed (Participants) | 30 | 31 | 30
  Day 22 to 28 | 1.93 (2.65) | 1.83 (2.55) | 1.45 (1.76)
  Day 29 to 35: number analyzed (Participants) | 31 | 32 | 31
  Day 29 to 35 | 1.76 (2.79) | 1.62 (2.17) | 1.53 (1.73)
  Day 36 to 42: number analyzed (Participants) | 32 | 30 | 31
  Day 36 to 42 | 1.86 (3.36) | 1.42 (1.65) | 1.59 (1.92)
  Day 43 to 49: number analyzed (Participants) | 33 | 31 | 28
  Day 43 to 49 | 1.85 (3.53) | 1.33 (1.44) | 1.71 (2.05)
  Day 50 to 56: number analyzed (Participants) | 33 | 30 | 28
  Day 50 to 56 | 2.16 (4.83) | 1.52 (1.94) | 1.87 (2.32)
  Day 57 to 63: number analyzed (Participants) | 32 | 29 | 30
  Day 57 to 63 | 2.59 (6.63) | 1.43 (1.73) | 1.54 (1.56)
  Day 64 to 70: number analyzed (Participants) | 30 | 30 | 30
  Day 64 to 70 | 2.69 (6.43) | 1.50 (1.76) | 1.48 (1.65)
  Day 71 to 77: number analyzed (Participants) | 28 | 27 | 30
  Day 71 to 77 | 1.69 (1.96) | 1.39 (1.84) | 1.48 (1.44)
  Day 78 to 84: number analyzed (Participants) | 29 | 30 | 31
  Day 78 to 84 | 1.27 (1.56) | 2.04 (3.11) | 1.47 (1.41)

9. Secondary Outcome: Number of Participants With Physician Global Assessment (PGA) at Day 42 and Day 84
Description: Physician Global Assessment (PGA) consisted of a single physician-rated question assessing participant's status as 'excellent', 'good', 'moderate', 'poor', 'worsening' or 'not applicable (NA)'. Number of participants were categorically summarized.
Time Frame: Days 42 and 84
Population: Evaluable population included participants who received any study drug and were followed according to the protocol through Day 42. Here, "Number Analyzed" signified those participants who were evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
Participants
  Day 42: Excellent: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Excellent | 9 | 10 | 10
  Day 42: Good: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Good | 12 | 19 | 16
  Day 42: Moderate: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Moderate | 8 | 3 | 7
  Day 42: Poor: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Poor | 3 | 3 | 2
  Day 42: Worsening: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Worsening | 1 | 1 | 0
  Day 42: Not applicable: number analyzed (Participants) | 34 | 36 | 36
  Day 42: Not applicable | 1 | 0 | 1
  Day 84: Excellent: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Excellent | 8 | 12 | 11
  Day 84: Good: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Good | 15 | 13 | 11
  Day 84: Moderate: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Moderate | 7 | 3 | 9
  Day 84: Poor: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Poor | 3 | 4 | 1
  Day 84: Worsening: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Worsening | 2 | 3 | 0
  Day 84: Not applicable: number analyzed (Participants) | 36 | 35 | 32
  Day 84: Not applicable | 1 | 0 | 0

10. Secondary Outcome: Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]) Scores
Description: Asthma Quality of Life Questionnaire (Standardized Version) (AQLQ[S]): a 32-item questionnaire that measures the functional impairments experienced by adult participants including 4 domains (symptoms, activity limitations, emotional function, and environmental stimuli). Participants were asked to recall their experiences during the previous 2 weeks and to score each of the 32 questions on a 7-point scale ranging from 7 (no impairment) to 1 (severe impairment). The overall score was calculated as the mean response to all questions. The 4 domain scores were the means of the responses to the questions in each of the domains. Overall AQLQ score and 4 domain scores ranged from 7 (no impairment) to 1 (severe impairment).
Time Frame: Days 0, 42, and 84
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
units on a scale
  Overall: Day 0 | 3.14 (0.91) | 3.18 (0.95) | 3.35 (1.11)
  Overall: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Overall: Day 42 | 4.74 (1.65) | 4.76 (1.46) | 5.16 (1.44)
  Overall: Day 84: number analyzed (Participants) | 35 | 35 | 32
  Overall: Day 84 | 4.91 (1.71) | 5.01 (1.44) | 5.11 (1.35)
  Symptoms: Day 0 | 2.84 (0.94) | 2.79 (1.08) | 3.11 (1.25)
  Symptoms: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Symptoms: Day 42 | 4.77 (1.82) | 4.82 (1.45) | 5.19 (1.62)
  Symptoms: Day 84: number analyzed (Participants) | 35 | 35 | 32
  Symptoms: Day 84 | 4.94 (1.68) | 4.95 (1.53) | 5.09 (1.36)
  Activity limitation: Day 0 | 3.56 (0.97) | 3.74 (1.13) | 3.98 (1.29)
  Activity limitation: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Activity limitation: Day 42 | 4.96 (1.54) | 4.92 (1.51) | 5.30 (1.42)
  Activity limitation: Day 84: number analyzed (Participants) | 35 | 35 | 32
  Activity limitation: Day 84 | 5.11 (1.74) | 5.23 (1.36) | 5.24 (1.44)
  Emotional function: Day 0: number analyzed (Participants) | 36 | 36 | 35
  Emotional function: Day 0 | 2.73 (1.25) | 2.44 (1.16) | 2.47 (1.48)
  Emotional function: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Emotional function: Day 42 | 4.30 (1.96) | 4.35 (1.77) | 4.91 (1.66)
  Emotional function: Day 84: number analyzed (Participants) | 35 | 35 | 32
  Emotional function: Day 84 | 4.59 (2.04) | 4.59 (1.75) | 4.84 (1.73)
  Environmental stimuli: Day 0 | 3.35 (1.31) | 3.72 (1.29) | 3.42 (1.48)
  Environmental stimuli: Day 42: number analyzed (Participants) | 33 | 36 | 36
  Environmental stimuli: Day 42 | 4.59 (1.69) | 4.63 (1.53) | 4.99 (1.44)
  Environmental stimuli: Day 84: number analyzed (Participants) | 34 | 35 | 32
  Environmental stimuli: Day 84 | 4.69 (1.80) | 5.08 (1.62) | 5.13 (1.35)

11. Secondary Outcome: Number of Healthcare Resources Utilized by Resource Type
Description: Healthcare resource use was summarized by resource type from information on asthma exacerbations, and asthma related medications. Healthcare resource utilization assessed the total number of hospitalizations, urgent care, primary care clinic visits, asthma specialist clinic visits, telephone calls, and home management.
Time Frame: Day 0 to Day 168
Population: as for outcome 1
Measure: Number; unit: healthcare resources
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36 | 36
healthcare resources
  Hospitalizations | 64 | 40 | 43
  Urgent care | 2 | 0 | 0
  Primary care clinic visits | 3 | 1 | 5
  Asthma specialist clinic visits | 5 | 5 | 0
  Telephone calls | 6 | 1 | 4
  Home management | 2 | 1 | 4

12. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) for Benralizumab
Description: The Cmax of benralizumab is reported. Non-compartmental pharmacokinetic (PK) analysis was used for evaluation.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: Safety population included all participants who received any study drug. Only participants in benralizumab arms were included in pharmacokinetic evaluation. Only those participants who had PK values above the quantification limit were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 32 | 33
microgram per milliliter (mcg/mL) | 7.03 (1.78) | 26.7 (6.49)

13. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Last Quantifiable Concentration (AUClast) for Benralizumab
Description: AUClast = area under the concentration-time curve from time 0 to last measurable concentration. Non-compartmental PK analysis was used for evaluation.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 31 | 27
microgram*day per milliliter | 65.7 (18.5) | 263 (64.1)

14. Secondary Outcome: Area Under the Serum Concentration-Time Curve From Time 0 to Extrapolated Infinite Time (AUC [0 - Infinity]) for Benralizumab
Description: AUC [0 - infinity] = Area under the serum concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - infinity). It is obtained from AUC (0 - t) plus AUC (t - infinity). Non-compartmental PK analysis was used for evaluation.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: microgram*day per milliliter
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 31 | 27
microgram*day per milliliter | 67.1 (18.0) | 268 (65.7)

15. Secondary Outcome: Systemic Clearance (CL) for Benralizumab
Description: Systemic clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Non-compartmental PK analysis was used for evaluation. Clearance was normalized to participant's body weight.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliliter per kilogram per day
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 31 | 27
milliliter per kilogram per day | 4.92 (1.96) | 3.97 (1.02)

16. Secondary Outcome: Terminal Phase Elimination Half-Life (t1/2) for Benralizumab
Description: Terminal phase elimination half-life is the time measured for the serum concentration to decrease by one half. Non-compartmental PK analysis was used for evaluation.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 31 | 27
days | 11.5 (3.14) | 13.2 (2.39)

17. Secondary Outcome: Volume of Distribution of the Central Compartment (Vc) for Benralizumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Vc = volume of distribution of the central compartment, calculated as Dose/Cmax; where Cmax = maximum observed serum concentration. Non-compartmental PK analysis was used for evaluation. Results were normalized to participant's body weight.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: milliliter per kilogram (mL/kg)
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 32 | 33
milliliter per kilogram (mL/kg) | 46.4 (17.0) | 39.8 (10.3)

18. Secondary Outcome: Volume of Distribution at Steady State (Vss) for Benralizumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired serum concentration of a drug. Vss = steady state volume of distribution, calculated as MRT*CL, where MRT is the Mean Residence Time and CL is systemic clearance; which is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Non-compartmental PK analysis was used for evaluation. Results were normalized to participant's body weight.
Time Frame: Predose and 1 hour post-end of infusion on Day 0; Days 7, 42, and 84
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 31 | 27
mL/kg | 71.8 (23.2) | 64.0 (15.1)

19. Secondary Outcome: Number of Participants With Anti-Drug Antibodies to Benralizumab
Description: Number of participants with anti-drug antibodies to benralizumab is reported.
Time Frame: Day 0 and 84
Population: Safety population included all participants who received any study drug. Only participants from benralizumab arms were included in immunogenicity evaluation. Only participants with adequate sample were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
Number analyzed (Participants) | 36 | 36
Participants
  Day 0: number analyzed (Participants) | 36 | 31
  Day 0 | 1 | 0
  Day 84: number analyzed (Participants) | 35 | 30
  Day 84 | 2 | 4

ADVERSE EVENTS:
Time Frame: Day 0 to Day 84
Arm/Group | Placebo | Benralizumab 0.3 mg/kg | Benralizumab 1.0 mg/kg
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/36 | 0/36
Serious Adverse Events (participants affected / at risk) | 9/38 | 8/36 | 11/36
Other Adverse Events (participants affected / at risk) | 28/38 | 30/36 | 28/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Benralizumab 0.3 mg/kg (N=36) | Benralizumab 1.0 mg/kg (N=36)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 9 (16) | 4 (8) | 6 (9)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=38) | Benralizumab 0.3 mg/kg (N=36) | Benralizumab 1.0 mg/kg (N=36)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Procedural nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 2 (2)
Feeling cold (General disorders) | 1 (1) | 1 (1) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site oedema (General disorders) | 0 (0) | 1 (1) | 0 (0)
Infusion site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Infusion site rash (General disorders) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (2) | 2 (2)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 3 (3) | 2 (2) | 2 (3)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Otitis externa (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Vaginitis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Ear injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1)
Skeletal injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Stab wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 3 (3)
Blood phosphorus decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Blood pressure decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Urine analysis abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Magnesium deficiency (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2) | 5 (5) | 3 (3)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 4 (5) | 5 (7) | 9 (10)
Hyposmia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (3)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 18 (36) | 12 (34) | 14 (24)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 6 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome. The PIs also agree for data to be presented first as a joint, multi-center publication.